CLINICAL TRIAL: NCT04131036
Title: Effects of Emicizumab vs. Factor VIII Prophylaxis on Joint and Bone Health in Severe Hemophilia A
Acronym: EmiMSK
Status: Recruiting | Type: Observational
Sponsor: Washington Institute for Coagulation (Other)
Collaborators: Genentech, Inc. (Industry)
Responsible Party: Principal Investigator, Rebecca Kruse-Jarres, MD, MPH, Executive/Medical Director, Washington Center for Bleeding Disorders at Washington Institute for Coagulation, Washington Institute for Coagulation
Other Study IDs: ML40714
Record Dates: First submitted 2019-10-14; First posted 2019-10-18 (Actual); Last update posted 2023-09-05 (Actual); Status verified 2023-08

CONDITIONS: Hemophilia A
Keywords: Hemophilia A; Joint Health; Bone Density; Emicizumab; factor VIII prophylaxis
MeSH Terms: conditions — Hemophilia A | interventions — Bone Density

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Biospecimen Retention: Samples With DNA — Plasma samples for biomarkers for storage in the data and sample research repository at Washington Institute for Coagulation
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm A: Male patients with severe Hemophilia A who use prophylaxis with IV factor VIII concentrate with intended trough >1%.
  Interventions: Other: assessment of joint health and bone density
- Arm B: Male patients with severe Hemophilia A who use prophylaxis with SQ emicizumab.
  Interventions: Other: assessment of joint health and bone density

INTERVENTIONS:
Other: assessment of joint health and bone density — We propose to study longitudinal joint and bone density changes in patients with severe Hemophilia A.

SUMMARY:
The investigators propose to study longitudinal joint and bone density changes in patients with severe Hemophilia A. Per current standard of care, most patients are on prophylactic FVIII replacement therapy intravenously several times weekly with a goal of keeping the trough >1% FVIII. Recent phase 3 data suggest superior bleed protection with emicizumab prophylaxis every 1-2 weeks. It is the purpose of this study to longitudinally assess joint health and bone density over 3 years and to compare the effect of routine factor VIII prophylaxis with emicizumab prophylaxis.

DETAILED DESCRIPTION:
Summary: This retrospective/prospective, non-randomized controlled study, whereby patients will be included in 1 of 2 groups depending on their current treatments as outlined below. Patients will be assigned to a specific group by the clinician/PI based on their current regimen with the intent to stay on this regimen for the next 3 years.

Duration of Study and Subject Participation: Study subject enrollment is anticipated to occur over about 12 months and study duration per subject will be 3 years. Thus a total study duration of 4 years is anticipated.

Intervention: By using musculoskeletal ultrasound, the investigators will measure joint health among participants and assess joint health changes over 3 years compared between group A (factor prophylaxis) vs. group B (emicizumab prophylaxis) as assessed by MSKUS at baseline and after 3 years. Other outcomes such as bone density, comparative assessment of joint and overall health status, and exploration of potential biomarkers for joint and bone health will also be assessed.

ELIGIBILITY:
Inclusion Criteria:

* Male gender
* Severe hemophilia A (factor VIII < 1%)
* Age ≥ 16 year
* Either on prophylaxis with factor VIII or emicizumab with the intention to stay on the current regimen for the next 3 years
* Willing and able to give written informed consent/assent
* Willing to undergo MSKUS, DEXA scan +/- collection of blood sampling for repository biomarkers
* Willing to come in for baseline and 3 yearly visits
* Willing to answer phone survey for bleeding and safety every 3 months

Exclusion Criteria:

* Current FVIII inhibitor of > 0.6 BU
* Unable to take FVIII replacement
* Other known bleeding disorder
* Other rheumatologic disorder affecting joints
* Other known neuromotor defect (making physical exam difficult)

Min Age: 16 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Male severe Hemophilia A patients at one of the several Hemophilia Treatment Center sites participating in this study and who meet the eligibility criteria and are interested in participating in the study.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2019-04-04 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
joint health comparison | 3 years
  Joint health changes over 3 years compared between group A (factor prophylaxis) vs. group B (emicizumab prophylaxis) as assessed by MSKUS at baseline and after 3 years.

SECONDARY OUTCOMES:
bone density comparison | 3 years
  Bone density changes over 3 years compared between group A (factor prophylaxis) vs. group B (emicizumab prophylaxis) as assessed by DEXA scan at baseline and after 3 years.
comparative assessment of joint and overall health | 3 years
  Observational comparative assessment of joint and overall health status evaluated by activity level, functional assessment, pain assessment, joint examination, and adherence.
mid-point assessment of joint health and bone density | 2 years
  Observational assessment of joint health and bone density at 1 and 2 years in the different groups.
biomarkers for joint and bone health | through completion of study, average 3 years
  Exploration of potential biomarkers for joint and bone health.

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca Kruse-Jarres, MD, MPH, Principal Investigator — Washington Institute for Coagulation
Locations (4):
- United States (4):
  - Orthopedic Hemophilia Treatment Center, Los Angeles, California
  - Hemophilia and Thrombosis Treatment Center, University of California, San Diego, San Diego, California
  - The University of Texas Health Science Center at San Antonio, San Antonio, Texas
  - Washington Center for Bleeding Disorders at Washington Institute for Coagulation, Seattle, Washington

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Forsyth AL, Giangrande P, Hay CR, Kenet G, Kessler CM, Knobl PN, Llinas A, Santagostino E, Young G. Difficult clinical challenges in haemophilia: international experiential perspectives. Haemophilia. 2012 Jul;18 Suppl 5:39-45. doi: 10.1111/j.1365-2516.2012.02887.x. PMID 22757683
- [Background] Manco-Johnson MJ, Abshire TC, Shapiro AD, Riske B, Hacker MR, Kilcoyne R, Ingram JD, Manco-Johnson ML, Funk S, Jacobson L, Valentino LA, Hoots WK, Buchanan GR, DiMichele D, Recht M, Brown D, Leissinger C, Bleak S, Cohen A, Mathew P, Matsunaga A, Medeiros D, Nugent D, Thomas GA, Thompson AA, McRedmond K, Soucie JM, Austin H, Evatt BL. Prophylaxis versus episodic treatment to prevent joint disease in boys with severe hemophilia. N Engl J Med. 2007 Aug 9;357(6):535-44. doi: 10.1056/NEJMoa067659. PMID 17687129
- [Background] Oldenburg J. Optimal treatment strategies for hemophilia: achievements and limitations of current prophylactic regimens. Blood. 2015 Mar 26;125(13):2038-44. doi: 10.1182/blood-2015-01-528414. Epub 2015 Feb 23. PMID 25712992
- [Background] Foltz V, Gandjbakhch F, Etchepare F, Rosenberg C, Tanguy ML, Rozenberg S, Bourgeois P, Fautrel B. Power Doppler ultrasound, but not low-field magnetic resonance imaging, predicts relapse and radiographic disease progression in rheumatoid arthritis patients with low levels of disease activity. Arthritis Rheum. 2012 Jan;64(1):67-76. doi: 10.1002/art.33312. PMID 21904998
- [Background] McAlindon TE, Bannuru RR. Osteoarthritis: Is viscosupplementation really so unsafe for knee OA? Nat Rev Rheumatol. 2012 Nov;8(11):635-6. doi: 10.1038/nrrheum.2012.152. Epub 2012 Sep 11. No abstract available. PMID 22964536
- [Background] Porta F, Gargani L, Kaloudi O, Schmidt WA, Picano E, Damjanov N, Matucci-Cerinic M. The new frontiers of ultrasound in the complex world of vasculitides and scleroderma. Rheumatology (Oxford). 2012 Dec;51 Suppl 7:vii26-30. doi: 10.1093/rheumatology/kes336. PMID 23230091
- [Background] Ceponis A, Wong-Sefidan I, Glass CS, von Drygalski A. Rapid musculoskeletal ultrasound for painful episodes in adult haemophilia patients. Haemophilia. 2013 Sep;19(5):790-8. doi: 10.1111/hae.12175. Epub 2013 May 15. PMID 23672827
- [Background] Kidder W, Nguyen S, Larios J, Bergstrom J, Ceponis A, von Drygalski A. Point-of-care musculoskeletal ultrasound is critical for the diagnosis of hemarthroses, inflammation and soft tissue abnormalities in adult patients with painful haemophilic arthropathy. Haemophilia. 2015 Jul;21(4):530-7. doi: 10.1111/hae.12637. Epub 2015 Jan 27. PMID 25623830
- [Background] Aznar JA, Perez-Alenda S, Jaca M, Garcia-Dasi M, Vila C, Moret A, Querol F, Bonanad S. Home-delivered ultrasound monitoring for home treatment of haemarthrosis in haemophilia A. Haemophilia. 2015 Mar;21(2):e147-e150. doi: 10.1111/hae.12622. Epub 2015 Jan 27. No abstract available. PMID 25623041
- [Background] Martinoli C, Della Casa Alberighi O, Di Minno G, Graziano E, Molinari AC, Pasta G, Russo G, Santagostino E, Tagliaferri A, Tagliafico A, Morfini M. Development and definition of a simplified scanning procedure and scoring method for Haemophilia Early Arthropathy Detection with Ultrasound (HEAD-US). Thromb Haemost. 2013 Jun;109(6):1170-9. doi: 10.1160/TH12-11-0874. Epub 2013 Apr 4. PMID 23571706
- [Background] Paschou SA, Anagnostis P, Karras S, Annweiler C, Vakalopoulou S, Garipidou V, Goulis DG. Bone mineral density in men and children with haemophilia A and B: a systematic review and meta-analysis. Osteoporos Int. 2014 Oct;25(10):2399-407. doi: 10.1007/s00198-014-2773-7. Epub 2014 Jul 8. PMID 25001982
- [Background] Kempton CL, Antoniucci DM, Rodriguez-Merchan EC. Bone health in persons with haemophilia. Haemophilia. 2015 Sep;21(5):568-77. doi: 10.1111/hae.12736. Epub 2015 Jul 14. PMID 26172840
- [Background] Liel MS, Greenberg DL, Recht M, Vanek C, Klein RF, Taylor JA. Decreased bone density and bone strength in a mouse model of severe factor VIII deficiency. Br J Haematol. 2012 Jul;158(1):140-3. doi: 10.1111/j.1365-2141.2012.09101.x. Epub 2012 Apr 2. No abstract available. PMID 22469061
- [Background] Lau AG, Sun J, Hannah WB, Livingston EW, Heymann D, Bateman TA, Monahan PE. Joint bleeding in factor VIII deficient mice causes an acute loss of trabecular bone and calcification of joint soft tissues which is prevented with aggressive factor replacement. Haemophilia. 2014 Sep;20(5):716-22. doi: 10.1111/hae.12399. Epub 2014 Apr 8. PMID 24712867
- [Background] Boban A, Zupancic Salek S, Kastelan D, Nemet D. Quantitative ultrasound and dual energy X-ray absorptiometry in the assessment of osteoporosis in patients with haemophilia. Haemophilia. 2014 Nov;20(6):e420-2. doi: 10.1111/hae.12529. No abstract available. PMID 25354773